CLINICAL TRIAL: NCT07330986
Title: Influenza A-associated Pulmonary Aspergillosis in Patients Admitted to the Intensive Care Unit in China: a Retrospective Cohort Study
Brief Title: Influenza A-associated Pulmonary Aspergillosis in Patients Admitted to the Intensive Care Unit in China
Status: Completed | Type: Observational
Sponsor: Jianfeng Xie (Other)
Responsible Party: Sponsor-Investigator, Jianfeng Xie, Professor, Southeast University, China
Organization: Southeast University, China (Other)
Other Study IDs: 2025ZDSYLL509-P01
Record Dates: First submitted 2025-12-05; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: ICU; Invasive Pulmonary Aspergillosis; Influenza A
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: IPA and non-IPA groups — Patients were divided into IPA and non-IPA groups according to FUNDICU criteria.

SUMMARY:
Invasive pulmonary aspergillosis (IPA) has traditionally been considered a disease of the severely immunocompromised host. However, emerging evidence over the past decade has identified severe influenza as a significant risk factor for IPA, termed influenza-associated pulmonary aspergillosis (IAPA) . The reported incidence of IAPA in ICU patients ranges from 11% to 32%, with associated mortality exceeding 50% in some cohorts.

The pathophysiology of IAPA is thought to involve influenza virus-induced damage to the respiratory epithelium, which impairs mucociliary clearance and disrupts local immune defenses, thereby facilitating invasion by aspergillus species. Studies from recent influenza seasons report IAPA incidences ranging from 16% to 23% in critically ill patients, with associated mortality rates soaring to over 50% . This mortality is substantially higher than that observed in influenza patients without IPA, underscoring the severity of this co-infection.

Despite this recognized threat, significant knowledge gaps remain. Existing studies on IAPA are predominantly single-center or include a limited number of patients, with considerable heterogeneity in their outcomes, constraining the generalizability of their findings . A comprehensive understanding of the specific risk factors that predispose influenza patients to IPA is crucial for early identification and intervention. Furthermore, the clinical course and determinants of mortality specifically within the IAPA population are not yet fully elucidated.

Therefore, we We conducted a retrospective, multicenter cohort study across 20 ICUs in China. Patients were categorized into IPA and non-IPA groups based on FUNDICU diagnostic criteria (clinical, radiological, and mycological evidence) to describe the risk factors, clinical characteristics and outcomes of critically ill patients with IAPA.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥18 years)
* patients admitted to the ICU between November 1, 2024, and February 28, 2025
* patients with acute respiratory failure due to laboratory-confirmed Influenza A pneumonia (defined by a positive PCR test on respiratory specimens)

Exclusion Criteria:

* patients with readmission to the ICU
* patients with incomplete clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the ICU between November 1, 2024, and February 28, 2025, with acute respiratory failure due to laboratory-confirmed Influenza A pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 542 (Actual)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
60-day mortality | From day 1 to day 60 after ICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Key Laboratory of Critical Care Medicine, Department of Critical Care Medicine, Zhongda Hospital, Southeast University, Nanjing, China